CLINICAL TRIAL: NCT04426136
Title: Qiang Sun，Department of Breast Surgery, Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College.
Brief Title: A Prospective Cohort Study Comparing Disparity in Surgical Procedure (Wide Local Excision Only vs Any Other Surgery Procedures) Among the Elderly Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-2020-EBC
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Elderly Patient; Wide Local Excision; Surgery; Survival Outcomes
Keywords: elderly; breast cancer; wide local excision; survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1. WLE group: patients in this group receiving WLE merely
- 2. other method group: patients in this group receiving any other surgical procedures except WLE

SUMMARY:
The incidence and mortality rates of breast cancer are still increasing in both developing and developed countries. The number of women ≥70 years who are affected by breast cancer (BC) worldwide is also on the increase. Based on the largest population and increasing aging, BC is also rapidly increasing among the elderly in China. According to the epidemiological profile data regarding BC in China, the second onset age peak of BC morbidity occurred after 70 years old and in 2020, the proportion of patients older than 65 is expected to exceed one-fifth and reach 27.0% by 2030. However, some controversies remain to be resolved due to the lack of high quality evidence. The tumor biological behavior, treatment choice and treatment tolerance among the elderly prominently differ from their young counterparts. Besides, they are rarely enrolled in large-scale randomized clinical trials or prospective cohort studies and the results are obtained mainly from retrospective studies. Also, frequent deviations from the standard guidelines lead to insufficient or excessive treatments, though the so-called standard guidelines are based on the clinicopathological characteristics and research findings among the younger BC patients. Studies focusing on the global population confirmed that the biological behavior of tumors among elderly patients was more favorable compared with younger patients but did not transform into survival benefits eventually. Numerous prospective, randomized trials have demonstrated that breast conserving surgery (BCS), consisting of segmental mastectomy and radiation treatment with or without axillary lymph node dissection (ALND), is equivalent to mastectomy in terms of overall survival (OS) and disease free survival (DFS) for patients with early stage breast carcinoma. Presentation of the ACOZOG-Z011 study results in 2011 resulted in a downward trend in the use of a completion axillary lymph node dissection in early breast cancer patients with 1-2 positive sentinel lymph nodes (SLN), treated with wide local excision (WLE) and whole breast irradiation. However, there is little evidence regarding the optimal axillary treatment in elderly breast cancer patients, since these patients are often excluded from clinical trials. We had done a retrospective study of breast cancer in the elderly, which demonstrated that those who with complex comorbidities receiving wide local excision merely were about 1.5 times more than those who without (71.2% vs 46.0%, p<0.001). However, it is paradoxical that, on the one hand, the risk of dying from breast cancer may increase if patients do not receive the standard treatment; on the other hand, they could not live long enough to benefit or even suffer more from the standard treatment. The key is to figure out who they are. Given the high proportion of patients treated only with WLE, we believe that it is important to compare the effects of different surgical procedures on prognosis among the elderly BC patient in a prospective cohort study, to be more specific, comparing the WLE versus any other surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer
* Received surgical treatment in this institution
* Specific surgical method data available
* Demographic and pathological data available
* No clear evidence of distant metastasis
* Agree to participate in the trial and receive long-term follow-up

Exclusion Criteria:

* Being intolerant of surgical treatment
* Distant metastases have been merged
* Patients who had simultaneous bilateral breast cancer
* Follow-up interval being less than 12 months except reaching endpoints of observation

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We intend to enroll all patients who have been treated in the breast surgery department of our hospital and meet the inclusion criteria from the date of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
disease free survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 72 months
  the time interval from surgery to disease recurrence or metastasis or considered as still alive at the observation deadline or missed during follow-up
overall survival | From date of surgery until the date of death from any cause, assessed up to 72 months
  the time interval from surgery to all cause death or considered as still alive at the observation deadline or missed during follow-up
breast cancer-specific survival | From date of surgery until the date of death from breast cancer related cause, assessed up to 72 months
  the time interval from surgery to breast cancer related death or considered as still alive at the observation deadline or missed during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Breast Surgery,Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided